CLINICAL TRIAL: NCT01595074
Title: The Identification, Validation and Implemention of Prognostic and/or Predictive Biomarkers for Adjuvant Chemotherapy in Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Biomarkers in Predicting Treatment Response in Samples From Patients With Early-Stage Non-Small Cell Lung Cancer Previously Treated With Adjuvant Chemotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2012-01965; LACE-BIO-2#1; CDR0000733532
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-08

CONDITIONS: Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

GROUPS / COHORTS (1):
- Ancillary-Correlative (laboratory biomarkre analysis): Archived RNA and DNA samples are analyzed for gene expression, mutations, and variations by RT-qPCR, MassARRAY, molecular inversion probe assay, and microarray assays. Results are then compared with patients' clinical outcomes.
  Interventions: Other: medical chart review; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: medical chart review — Correlative studies
  Other Names: chart review
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in predicting treatment response in samples from patients with early-stage non-small cell lung cancer previously treated with adjuvant chemotherapy. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Validation of the 15-gene prognostic and predictive messenger (m) ribonucleic acid (RNA) signature on Lung Adjuvant Cisplatin Evaluation (LACE)-Bio formalin-fixed, paraffin-embedded tissue (FFPE) tumor samples.

II. Exploratory evaluation of the prognostic and predictive values of known potential oncogenic mutations using LACE-Bio FFPE tumor samples.

III. Exploratory evaluation of the prognostic and predictive values of gene copy variations using LACE-Bio FFPE tumor samples.

IV. Exploratory identification and evaluation of prognostic and predictive value of novel genomic aberrations discovered by Next Generation Sequencing on LACE-Bio tumor samples.

OUTLINE:

Archived RNA and DNA samples are analyzed for gene expression, mutations, and variations by reverse transcriptase (RT)-polymerase chain reaction (qPCR), mass spectrometry (MassARRAY), molecular inversion probe assay, and microarray assays. Results are then compared with patients' clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients treated in 4 adjuvant chemotherapy (ACT) for early-stage non-small cell lung cancer (NSCLC) pivotal trials:

  * International Adjuvant Lung Cancer Trail (IALT)
  * Cancer and Leukemia Group B (CALGB)-9633
  * CAN-NCIC-BR10
  * Adjuvant Navelbine International Trialist Association (ANITA)
* Not specified
* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2012-05; Primary Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the 15-gene prognostic and predictive mRNA signature by quantitative Nuclease Protection Assay (qNPA) assay and NanoString assay | Post-RNA extraction from tissue
Prognostic and predictive value of known potential oncogenic mutations and gene copy variations of novel genomic aberrations on disease free survival (DFS) and overall survival (OS) | Post-RNA extraction from tissue
  Survival curves will be estimated using Kaplan-Meier methods and compared with the log-rank test. The hypothesis of constant risk ratio over time in the Cox proportional hazards (PH) model will be tested by introducing a time-dependent interaction with the marker or using Schoenfeld's residuals.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Seymour, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada